CLINICAL TRIAL: NCT00005965
Title: Phase II Clinical Trial of Bryostatin-1, NSC 339555, and Cisplatin in Patients With Recurrent and/or Advanced Inoperable Squamous Cell, Adeno or Adenosquamous Cell Carcinoma of the Cervix
Brief Title: Bryostatin-1 Plus Cisplatin in Treating Patients With Recurrent or Advanced Cancer of the Cervix
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: MTS-99-1113-ME; CDR0000067948 (Registry Identifier: PDQ (Physician Data Query)); NCI-T99-0082
Record Dates: First submitted 2000-07-05; First posted 2004-03-05 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2004-07

CONDITIONS: Cervical Cancer
Keywords: stage III cervical cancer; recurrent cervical cancer; stage IVB cervical cancer; stage IVA cervical cancer; cervical squamous cell carcinoma; cervical adenocarcinoma; cervical adenosquamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — bryostatin 1; Cisplatin

INTERVENTIONS:
Drug: bryostatin 1
Drug: cisplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of bryostatin-1 plus cisplatin in treating patients who have recurrent or advanced cancer of the cervix.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and efficacy of bryostatin-1 plus cisplatin in patients with recurrent or advanced carcinoma of the cervix. II. Determine the response rate, progression free interval, and duration of survival of these patients when treated with this regimen.

OUTLINE: This is a multicenter study. Patients receive bryostatin-1 IV over 1 hour and cisplatin IV over 1 hour on day 1. Treatment continues every 21 days in the absence of disease progression or unacceptable toxicity. Patients are followed until death.

PROJECTED ACCRUAL: A total of 37 patients will be accrued for this study over 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent or advanced carcinoma of the cervix not amenable to surgery or radiotherapy Squamous cell OR Adenocarcinoma OR Adenosquamous carcinoma Measurable disease Brain metastases treated with surgery or radiotherapy allowed if no residual symptoms or medications (e.g., anticonvulsants, corticosteroids)

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin greater than 9 g/dL Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) AST/ALT less than 2.5 times ULN Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No severe cardiac dysfunction or arrhythmia Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No concurrent unstable medical illness, infection, or other significant medical problem No clinically apparent neuropathy, including hearing loss No psychological, familial, sociological, or geographical conditions that may preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Prior neoadjuvant chemosensitization therapy allowed At least 3 weeks since prior chemotherapy (6 weeks since prior mitomycin or nitrosoureas) and recovered Prior cisplatin therapy allowed No prior chemotherapy for advanced disease Endocrine therapy: No concurrent corticosteroids Radiotherapy: At least 2 weeks since prior radiotherapy and recovered Surgery: Prior surgery allowed Other: No concurrent anticonvulsants No concurrent antiarrhythmic medication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farr R. Nezhat, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (6):
- United States (6):
  - Saint Vincent Catholic Medical Center of New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York

REFERENCES:
- [Result] Nezhat F, Wadler S, Muggia F, Mandeli J, Goldberg G, Rahaman J, Runowicz C, Murgo AJ, Gardner GJ. Phase II trial of the combination of bryostatin-1 and cisplatin in advanced or recurrent carcinoma of the cervix: a New York Gynecologic Oncology Group study. Gynecol Oncol. 2004 Apr;93(1):144-8. doi: 10.1016/j.ygyno.2003.12.021. PMID 15047228